CLINICAL TRIAL: NCT00766857
Title: The Effect of Exenatide Compared to Insulin Glargine on Cardiac Function and Metabolism in Type 2 Diabetic Patients With Congestive Heart Failure: a Randomized Comparator-controlled Trial
Brief Title: Effects of Exenatide in Type 2 Diabetic Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.H.H. Kramer, MD, PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC2008exe001; EudraCT: 2008-005325-10
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes Mellitus; Congestive Heart Failure
Keywords: Exenatide; Type 2 diabetes mellitus; Congestive heart failure; Incretin hormones; GLP-1 agonist; Cardiac metabolism; Insulin resistance; Cardiac MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Insulin Resistance | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Exenatide (Experimental)
  Interventions: Drug: exenatide
- 2. Insulin glargine (Active Comparator)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: exenatide — Exenatide 5 mcg BID for 4 weeks, subsequently increased to 10 mcg BID for the remainder of the study (total of 26 weeks).
  Other Names: exenatide-Byetta
  Arms: 1. Exenatide
Drug: Insulin glargine — Insulin glargine will be initiated at 10 IU QD, titrated according to fasting blood glucose concentrations based on general protocol-defined guidance.
  Other Names: insulin glargine-Lantus
  Arms: 2. Insulin glargine

SUMMARY:
The purpose of this study is to determine if exenatide will improve global cardiac function in patients with type 2 diabetes mellitus and congestive heart failure, by favorable effects on cardiac metabolism leading to improvement of cardiac efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Male and postmenopausal female
* Age 18 years an above
* Metformin therapy (stable, maximum tolerable dose for 2 months)
* HbA1c 6.5-10%
* Confirmed congestive heart failure (NHYA functional class II-IV)
* Ejection fraction < 50%
* Patients should receive a stable standard therapy for their cardiac condition for 3 months prior entering the study

Exclusion Criteria:

* Type 1 diabetes mellitus
* Serious renal or liver impairment
* (Receiving treatment for) malignant disease
* Cardiovascular event < 3 months prior to inclusion
* Acute congestive heart failure
* Any reason for not being able to sustain the imaging studies
* Pacemaker/ICD
* Contraindications for the use of exenatide/ insulin
* Use of insulin, thiazolidinediones, incretin-based therapies within 4 months of screening
* Chronic use of glucocorticoids, NSAIDs or centrally acting drugs (> 2 weeks) within 2 weeks immediately prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Magnetic Resonance (CMR) will be used to assess global cardiac function (LV ejection fraction). | week -2 and week 11

SECONDARY OUTCOMES:
Cardiac oxygen consumption, cardiac efficiency and stress perfusion will be assessed by Positron Emission Tomography (PET) using 11C-acetate and H2-15O | week -2 and week 26
Cardiac function, dimensions and scarring will be measured bij CMR | week -2 and week 26
Myocardial diastolic function parameters will be obtained bij trans thoracal echocardiography. Comparisons will be made of strain and torsion measures obtained bij CMR and echocardiography. | week -2 and week 26
Exercise capacity and performance will be assessed by a 6-minute walking test | week -1 and week 27

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Diamant, MD, PhD, Principal Investigator — VUMC Diabetes Center
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Chen WJY, Diamant M, de Boer K, Harms HJ, Robbers LFHJ, van Rossum AC, Kramer MHH, Lammertsma AA, Knaapen P. Effects of exenatide on cardiac function, perfusion, and energetics in type 2 diabetic patients with cardiomyopathy: a randomized controlled trial against insulin glargine. Cardiovasc Diabetol. 2017 May 19;16(1):67. doi: 10.1186/s12933-017-0549-z. PMID 28526033